CLINICAL TRIAL: NCT06955975
Title: The Effect of Pectin Supplementation on Geriatric With Frailty: A Randomised Placebo-Controlled Dietary Intervention Study
Acronym: GEOFF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Ana Valdes, Professor in Genetic and Molecular Epidemiology, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FMHS 280-0924
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Frailty at Older Adults; Pre-Frailty; Frailty; Diet; Dietary Fiber; Systemic Inflammatory Response
Keywords: Pectin; LM Pectin; Frailty; Pre-Frailty; Systemic inflammation; Dietary intervention; Gut microbiome
MeSH Terms: conditions — Frailty | interventions — Pectins; Whey Proteins

STUDY DESIGN:
Intervention Model Description: Controlled intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pectin (Active Comparator): 10g of pectin with 10g of whey protein and 10g of cocoa powder added as flavour will be provided to participants for 4 weeks.
  Interventions: Dietary Supplement: Pectin
- Whey protein (Placebo Comparator): 10g of whey protein with 10g of cocoa powder added as flavour will be provided to participants for 4 weeks.
  Interventions: Other: Whey protein

INTERVENTIONS:
Dietary Supplement: Pectin — 10g of pectin with 10g of whey protein and 10g of cocoa powder added as flavour were randomly allocated to eligible participants in order to test specific effects on gut microbiome composition and metabolic markers.
  Arms: Pectin
Other: Whey protein — 10g of whey protein with 10g of cocoa powder added as flavour served as the control/ placebo to compare the effects observed with pectin.
  Arms: Whey protein

SUMMARY:
The study involves the intake of Low-methoxy (LM) pectin (polysaccharides extracted from citrus peels), which are commonly found in the UK diet (not pharmacological agents), to test their effects on systematic inflammation in the body and gut microbiome composition. Study subjects will be healthy elderly with early signs of frailty or pre-frailty from the local population and will be asked to attend the laboratory on 2 occasions; before and after 4-week' supplementing the diet daily with either 10g of pectin with 10g of whey protein and 10g of cocoa powder added as flavour (active arm) or 10g of whey protein with 10g of cocoa powder added as flavour (placebo). Participants will be given the blinded products portioned in individual sachets, with instructions to add the contents of one sachet a day to 150ml of milk and to consume immediately.

At each study visit (~90 minutes), participants will be asked to provide a stool and blood sample, will have blood pressure, heart rate, weight, height, and waist/hip ratio measured, research team will perform physical functioning test (Time up and go test, 30-second sit to stand test) as well as participants will complete the quality-of-life questionnaire (SF-36), the Depression and Anxiety (HADS) and the Gastrointestinal Symptom Rating Scale (GSRS).

DETAILED DESCRIPTION:
The overall aim of the proposed project is to study the effect of daily ingestion of a dietary fibre (LM pectin) among frail population on anti-inflammatory and cardioprotective metabolic measures and to determine whether effects are mediated via the modulation of the gut microbiome and SCFAs production.

Specific Aim 1: To determine the effects of 4-weeks' pectin dietary supplementation on gut microbiome composition and diversity and the concentration of markers of intestinal permeability in the blood.

Specific Aim 2: To investigate the impact of daily pectin intake on physical functioning and subjective quality of life.

Specific Aim 3: To investigate the consequences of 4-weeks' daily ingestion of pectin on subjective measures of depression and anxiety among frail participants.

30 healthy elderly with early signs of frailty or pre-frailty will be recruited following a successful medical screening.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Participant eligibility includes those aged >65 years who have a body mass index (BMI) between 18.5 and 39.9 kg/m2.
* Participants who are considered as pre-frail or frail based on FRAIL (Simple Frailty Questionnaire).

Exclusion Criteria:

* Have gastrointestinal conditions e.g. malabsorptive conditions such as IBS/IBD, coeliac or functional conditions such as gastroparesis or food intolerances etc.
* History of major surgery which potentially limit participation or completion of the study.
* History of gastrointestinal resection surgery, including bariatric surgery.
* Used of antibiotics, antifungal medications, probiotics or prebiotics 90 days before the start of the study.
* Are taking the following medications: immunosuppressants, amiodarone and/or perhexiline.
* Are currently following or anticipated to commence a specialised commercially available weight loss diet and/or program.
* History of side effects towards probiotics or prebiotics.
* History or current psychiatric illness.
* History or current neurological condition (e.g. epilepsy).
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in microbiome profile | 4 weeks
  Change in microbiome profile, assessed using 16s RNA sequencing analysis of faecal samples provided pre and post the 4-week intervention period.
Change in inflammatory profile | 4 weeks
  Change in circulating markers of inflammation measured by ELISAs in serum samples collected pre and post the 4-week intervention period.
Changes in short chain fatty acids (SCFAs) | 4 weeks
  Change in serum SCFAs measured by mass spectrometry pre and post the 4-week intervention period.

SECONDARY OUTCOMES:
Change in systolic blood pressure (lying to standing) pre intervention | 4 minutes
  Change in systolic blood pressure (measured after 3 minutes of lying down and after 1 minute of standing), at pre-intervention study visit.
Change in systolic blood pressure (lying to standing) post intervention | 4 minutes
  Change in systolic blood pressure (measured after 3 minutes of lying down and after 1 minute of standing), at post-intervention study visit
Change in diastolic blood pressure (lying to standing) pre intervention | 4 minutes
  Change in diastolic blood pressure (measured after 3 minutes of lying down and after 1 minute of standing), at pre-intervention study visit.
Change in diastolic blood pressure (lying to standing) post intervention | 4 minutes
  Change in diastolic blood pressure (measured after 3 minutes of lying down and after 1 minute of standing), at post-intervention study visit.
Change in body mass index (BMI) | 4 weeks
  Change in BMI pre and post the 4-week intervention period.
Change in waist-to-hip ratio (WHR) | 4 weeks
  Change in WHR pre and post the 4-week intervention period.
Change in time up and go test (TUG) | 4 weeks
  Change in TUG pre and post the 4-week intervention period.
Change in 30-second sit to stand test | 4 weeks
  Change in 30-second sit to stand test pre and post the 4-week intervention period.
Change in Hospital Anxiety and Depression Score (HADS) | 4 weeks
  Change in anxiety score (min score 0, max 3 with higher score indicating higher anxiety like symptoms), and depression score (min 3, max 0 with lower the scores indicating higher depression like symptoms) measured pre and post the 4-week intervention.
Change in 36-Item Short Form Survey (SF-36) Questionnaire | 4 weeks
  Change in SF-36 scores pre and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Ana Valdes, PhD student candidate, Principal Investigator — University of Nottingham; Noor K Al-Tameemi, PhD student candidate, Study Director — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The research team will try their best to share statistical plan with other researchers